CLINICAL TRIAL: NCT01089985
Title: Use of Autologous Serum Eye-drops as Tears in Patients With Recalcitrant Dry Eye
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Singapore National Eye Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R724/08/2010
Record Dates: First submitted 2010-03-16; First posted 2010-03-19 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Xerophthalmia
MeSH Terms: conditions — Xerophthalmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Serum eye drops (Experimental): Patient's autologous serum is diluted in saline solution
  Interventions: Drug: Autologous serum eyedrops

INTERVENTIONS:
Drug: Autologous serum eyedrops — 3 times a day for the duration of the study

SUMMARY:
The purpose of this study is to examine the efficacy and safety of autologous serum eye drops in people with recalcitrant dry eye.

DETAILED DESCRIPTION:
A group of selected dry eye patients from the Singapore National Eye Centre who have exhausted the usual treatment options (lubricants, topical immunosuppressive and punctal occlusion) and not keen for tarsorrhaphy will be recruited. After informed consent, they will undergo plasmapheresis and start on daily autologous serum eyedrops for a period of 4 months. Clinical monitoring for standard dry eye parameters such as punctate corneal keratitis, Schirmers testing, tear break up time as well as severity and frequency of dry eye symptoms will be conducted. Tear inflammatory proteins captured on Schirmers paper pre and post treatment will be analysed as well.

ELIGIBILITY:
Inclusion Criteria:

* Seen at the dry eye service at the Singapore National Eye Centre
* Age between 21 and 75 years old
* Symptomatic for dry eye or VA worse than 6/12 in Snellen chart
* Presence of corneal punctate staining involving central zone
* Exhausted what is considered as standard therapy or therapy that is acceptable to the patient and the physician
* No contraindication for blood extraction/plasmapheresis

Exclusion Criteria:

* HIV/HCV/HBV/syphilis

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Staining | 4 months
  Grading of punctate corneal staining in the worse eye (second visit relative to first visit)

SECONDARY OUTCOMES:
Symptoms | 4 months
  The change in Visual Analog Score (Schaumberg D et al Ocular Surface 2009). The global score is calculated from 2 scores, the frequency and severity of dry eye symptoms.
  From .
Tear-production | 4 months
  Schirmers test result
Tear-proteins | 4 months
  Tear protein analysis
Tear-stability | 4 months
  Tear break up time
Cornea | 4 months
  other corneal findings such as scarring, vascularisation, filaments etc
Conjunctiva | 4 months
  Documentation of conjunctival hyperemia, chemosis, scarring

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, FRCS, MD, Principal Investigator — Singapore National Eye Centre; Ronald Chung, Principal Investigator — Singapore National Eye Centre; Roger Beuerman, Study Director — Singapore Eye Research Institute; Mickey Koh, Study Chair — Singapore General Hospital; Samanthila Waduthantri, Study Chair — Singapore National Eye Centre; Heng Joo Ng, Study Chair — Singapore General Hospital; Rohani Salleh, Study Chair — Singapore General Hospital
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore, Singapore